CLINICAL TRIAL: NCT05882760
Title: Comparison of Postoperative Sensitivity Following Placement with Different Restorative Materials in Vital Posterior Teeth
Brief Title: Postoperative Sensitivity Following Placement with Different Restorative Materials in Vital Posterior Teeth
Acronym: GCP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Responsible Party: Principal Investigator, Sarang Suresh, FCPS Trainee, Liaquat University of Medical & Health Sciences
Allocation: Not Applicable | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LUMHS/REC/-29
Record Dates: First submitted 2023-05-20; First posted 2023-05-31 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Sensitivity, Tooth
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Tetric N Bond Universal® (Experimental): Cavities in this group will be restored with Conventional Hybrid Composite Restoration bonded with Etch & Rinse Technique using Tetric N Bond Universal®.
  Interventions: Drug: Tetric N Bond Universal®
- Self Etch Tetric N Bond Universal® (Active Comparator): Cavities in this group will be restored with Conventional Hybrid Composite Restoration bonded with Self Etch Technique using Tetric N Bond Universal®.
  Interventions: Drug: Self Etch Tetric N Bond Universal®
- GC Fuji IX, GC, Japan® (Active Comparator): Cavities in this group will be restored with GC Fuji IX, GC, Japan®
  Interventions: Drug: GC Fuji IX, GC, Japan®
- Activa TM Bioactive Restorative ® (Active Comparator): Cavities in this group will be restored with Activa TM Bioactive Restorative ®
  Interventions: Drug: Activa TM Bioactive Restorative ®

INTERVENTIONS:
Drug: Tetric N Bond Universal® — Cavities will be restored with Conventional Hybrid Composite Restoration bonded with Etch & Rinse Tetric - N - Bond (Ivoclar)
  Arms: Tetric N Bond Universal®
Drug: Self Etch Tetric N Bond Universal® — Cavities will be restored with Conventional Hybrid Composite Restoration bonded with Self Etch Tetric N Bond Universal®
  Arms: Self Etch Tetric N Bond Universal®
Drug: GC Fuji IX, GC, Japan® — Cavities will be restored with GC Fuji IX, GC, Japan®
  Arms: GC Fuji IX, GC, Japan®
Drug: Activa TM Bioactive Restorative ® — Cavities will be restored with Activa TM Bioactive Restorative ®
  Arms: Activa TM Bioactive Restorative ®

SUMMARY:
There is a lack of long-term clinical studies comparing different restorative materials; most of the available studies have only looked at class I cavities or examined post-operative sensitivity in non-caries cervical lesions. The purpose of this study is to measure postoperative sensitivity in clinical settings at 3-month intervals for class 1 and 2 direct posterior restoration

ELIGIBILITY:
Inclusion Criteria:

Either gender Minimum age 18 years, maximum age 40 years. Class I & II Cavity on maxillary and mandibular 1st and 2nd molars. Vital maxillary and mandibular molar teeth that had occlusal contact with antagonist teeth.

Exclusion Criteria:

Irreversible Pulpitis diagnosed clinically and radiographically. Class I & Class II cavity of premolars and third molars Patients taking analgesic prior to treatment. History of allergic reaction to any dental material used in the study. History of parafunctional habits (bruxism and/or clenching) Malocclusion

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Post Operative Sensitivity | 3 Months
  Sensitivity will be recorded as present when a patient experienced more pain when the cold stimulus is applied on the restored tooth than on the control tooth is assessed using the modified visual analogue scale to any stimulus (occlusal function, cold/hot water, or sweets) every day by the patient until 7 days, then by the clinician on 7 days, 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Priya Rani, BDS, Principal Investigator — Liaquat University of Medical and Health Science
Locations (1):
- Institute of Dentistry, Liaquat University of Medical and Health Sciences, Hyderābād, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No